CLINICAL TRIAL: NCT03559335
Title: WBC Count, CRP, PCT, Neutrophil CD64 and Monocyte Human Leukocyte Antigen- DR Expression in the Diagnosis of Postoperative Infectious Complications in Colorectal Cancer Surgery
Brief Title: Inflammation Biomarkers in the Diagnosis of Postoperative Infectious Complications in Colorectal Cancer Surgery
Status: Completed | Type: Observational
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Principal Investigator, Achkasov Sergey, Professor Sc.State Scientific Centre of Coloproctology, Head of Surgical department of sugery and oncology of colon, Moscow,Russian Federation, State Scientific Centre of Coloproctology, Russian Federation
Other Study IDs: 79
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Biomarkers; Neutrophil CD64; Monocyte Human Leukocyte Antigen - DR; Postoperative Infectious Complications; C-reactive protein (CRP); Procalcitonin (PCT)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients after colorectal cancer surgery

SUMMARY:
This is a longitudinal, single-center, prospective study to determine the efficiency of WBC Count, CRP, PCT, Neutrophil CD64 and Monocyte Human Leukocyte Antigen- DR in the diagnosis of postoperative infectious complications in colorectal cancer surgery

DETAILED DESCRIPTION:
Blood samples for inflammation markers are carried out from patients with сolorectal cancer surgery in a single center on the day of the surgery in the operating room before intravenous fluid application started. Each patient receives systemic antibiotic prophylaxis for gramnegative and anaerobic bacteria on induction of anesthesia and prior to skin incision. A standardized protocol for general and epidural anesthesia is used. Values of WBC count, CRP, PCT, CD64n and HLA-DR monocyte are recorded before surgery and after surgery on POD (postoperative day) 1, 3 and 6 or 7. SIRS criteria on POD 1, 3, 6 or 7 and postoperative infections up to 30 days after surgery are recorded. SSIs (incisional, organ / space), pneumonia, central venous catheter related bloodstream infections (CRBSIs), urinary tract infections (UTIs) and enterocolitis records are taken. Microbial cultures are using as the gold standard. Criteria for SIRS reconsidered in the year 2001 by SCCM / ESICM / ACCP / ATS / SIS International Sepsis Definitions Conference and criteria for Dosage Control and Prevention (CDC) are taken into consideration. After discharge, each patient is being monitored by outpatient clinic examinations. The study will recruit approximately 100 patients during three consecutive years.

ELIGIBILITY:
Inclusion Criteria:

* Have a elective colorectal resection for colorectal cancer
* Have signed approved informed consent form for the study

Exclusion Criteria:

* Significant simultaneous surgical procedure (e.g., liver resection of metastasis)
* Bacterial infection at the time of surgery or antimicrobial therapy up to 4 weeks before surgery
* Neo-adjuvant chemotherapy and/or radiotherapy
* Autoimmune conditions
* Inflammatory bowel diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancer who undergo colorectal surgery at State Scientific Center of Coloproctology.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Postoperative inflammatory complications | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- State Scientific Centre of Coloproctology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Achkasov SI, Sukhina MA, Sushkov OI, Nabiev EN, Shakhmatov DG, Tarasov MA, Moskalev AI. [The role of neutrophil CD64 index in the diagnosis of infectious complications after colorectal resection]. Khirurgiia (Mosk). 2020;(10):29-35. doi: 10.17116/hirurgia202010129. Russian. PMID 33047583